CLINICAL TRIAL: NCT05190731
Title: Alterations in Bioelectric Activity at Acupuncture Jing-Well (Ting) Points Following CV4 Cranial Manipulation
Brief Title: Alterations in Bioelectric Activity at Acupuncture Points Following CV4 Cranial Manipulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jan T Hendryx (Other)
Responsible Party: Sponsor-Investigator, Jan T Hendryx, Clinical Professor of OPP and Family Medicine, Lake Erie College of Osteopathic Medicine
Organization: Lake Erie College of Osteopathic Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 24-177
Record Dates: First submitted 2021-12-29; First posted 2022-01-13 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Autonomic Imbalance
MeSH Terms: interventions — salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: Participants randomized to sham group or osteopathic cranial manipulative medicine treatment group
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Contact touch at occipital region, but no actual cranial manipulation (Sham Comparator): Each subject was treated with Sham by CSPOMM and NMM board-certified osteopathic physicians. The physician's finger pads of both hands were placed underneath the supine subject's head in contact on the occipital squama medial to the lambdoidal and occipitomastoid sutures. The subject's head rested passively on the finger pads for 3 minutes. No cranial manipulative forces were applied.
  Interventions: Other: Sham
- Osteopathic cranial manipulative medicine (Active Comparator): Each subject was treated with CV4 technique by CSPOMM and NMM board-certified osteopathic physicians. All CV4 treatments were performed by one individual according to standardized protocol. The physician's hands were placed underneath the occiput with the thenar eminences in contact on the occipital squama medial to the lambdoidal and occipitomastoid sutures. Inherent cranial rhythmic motion was identified and thenar eminences followed occipital motion anteriorly during the extension phase until a still point was attained. This position was held until the still point released (usually about 3 minutes) and normal cranial motion ensued.
  Interventions: Other: Osteopathic cranial manipulative medicine

INTERVENTIONS:
Other: Osteopathic cranial manipulative medicine — Osteopathic cranial manipulative medicine technique using compression of 4th ventricle technique
  Arms: Osteopathic cranial manipulative medicine
Other: Sham — Touch only, no osteopathic cranial manipulation
  Arms: Contact touch at occipital region, but no actual cranial manipulation

SUMMARY:
By measuring specific electrical parameters at acupuncture points that have been shown to correlate with ANS activity, the objectives of this study were to: 1) determine if CV4 has any influence on the bioelectric properties of the acupuncture meridian system, and 2) determine if CV4 affects the ANS.

DETAILED DESCRIPTION:
This study is designed to measure bioelectrical activity at acupuncture Ting (Jing-Well) points immediately before and after employing a specific Osteopathic Cranial Manipulative Medicine (OCMM) technique called CV4 (Compression of the 4th Ventricle) vs. a Sham treatment.

Ting (Jing-Well) points are acupuncture points located at the proximal edges of the finger- and toenails that represent the beginning and end of 14 acupuncture meridians as described in Traditional Chinese Medicine and Japanese systems. Measurement of electrical activity at Ting points is performed by a physicist who has extensive experience using a device known as the Apparatus for Meridian Identification (AMI). Data collected and analyzed by the AMI for both CV4 and Sham groups is compared statistically for significant differences in before vs. after electrical activity and specific acupuncture meridians affected. One particular analysis of After Polarization (AP) potentials correlates with changes in autonomic nervous system activity.

ELIGIBILITY:
Inclusion Criteria:

* Males and females from the Erie, PA, area aged 18-78 years
* Recruited by local flyers and word of mouth marketing
* Able to lay supine for about 30 minutes

Exclusion Criteria:

* Persons under the age of 18 years and persons unable to attend the in-person research sessions in Erie, PA.
* Identifiable acute illness of any kind
* Past medical history of stroke or transient ischemic attack within past 6 months
* Past medical history of intracranial hemorrhage, increased intracranial pressure, or seizure disorder
* Pregnant females

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2017-11-10 (Actual); Primary Completion 2018-06-24 (Actual); Study Completion 2018-11-07 (Actual)

PRIMARY OUTCOMES:
Autonomic Nervous System Activity at Acupuncture Ting Points | Within 15 minutes of sham or intervention
  Bioelectric skin conductance at acupuncture points

CONTACTS AND LOCATIONS:
Overall Officials: Jan Hendryx, DO, Principal Investigator — Lake Erie College of Osteopathic Medicine
Locations (1):
- LECOM Health, Erie, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data underlying the results appearing in a scientific publication after de-identification including text, table, figures and appendices.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data requests can be submitted beginning 9 months after article publication and data will remain accessible for up to 24 months thereafter. Extensions will be considered on a case-by-case basis.
Access Criteria: Please contact Director of Research, Lake Erie College of Osteopathic Medicine, 1858 West Grandview Blvd., Erie, PA, 16509

REFERENCES:
- [Background] Jakel A, von Hauenschild P. Therapeutic effects of cranial osteopathic manipulative medicine: a systematic review. J Am Osteopath Assoc. 2011 Dec;111(12):685-93. PMID 22182954
- [Background] Zurowska A, Malak R, Kolcz-Trzesicka A, Samborski W, Paprocka-Borowicz M. Compression of the Fourth Ventricle Using a Craniosacral Osteopathic Technique: A Systematic Review of the Clinical Evidence. Evid Based Complement Alternat Med. 2017;2017:2974962. doi: 10.1155/2017/2974962. Epub 2017 Oct 18. PMID 29234380
- [Background] Curi ACC, Maior Alves AS, Silva JG. Cardiac autonomic response after cranial technique of the fourth ventricle (cv4) compression in systemic hypertensive subjects. J Bodyw Mov Ther. 2018 Jul;22(3):666-672. doi: 10.1016/j.jbmt.2017.11.013. Epub 2017 Dec 9. PMID 30100295
- [Background] Abenavoli A, Badi F, Barbieri M, Bianchi M, Biglione G, Dealessi C, Grandini M, Lavazza C, Mapelli L, Milano V, Monti L, Seppia S, Tresoldi M, Maggiani A. Cranial osteopathic treatment and stress-related effects on autonomic nervous system measured by salivary markers: A pilot study. J Bodyw Mov Ther. 2020 Oct;24(4):215-221. doi: 10.1016/j.jbmt.2020.07.017. Epub 2020 Aug 4. PMID 33218514
- [Background] Arienti C, Farinola F, Ratti S, Dacco S, Fasulo L. Variations of HRV and skin conductance reveal the influence of CV4 and Rib Raising techniques on autonomic balance: A randomized controlled clinical trial. J Bodyw Mov Ther. 2020 Oct;24(4):395-401. doi: 10.1016/j.jbmt.2020.07.002. Epub 2020 Jul 31. PMID 33218540
- [Background] Rechberger V, Biberschick M, Porthun J. Effectiveness of an osteopathic treatment on the autonomic nervous system: a systematic review of the literature. Eur J Med Res. 2019 Oct 25;24(1):36. doi: 10.1186/s40001-019-0394-5. PMID 31653268
- [Background] Cutler MJ, Holland BS, Stupski BA, Gamber RG, Smith ML. Cranial manipulation can alter sleep latency and sympathetic nerve activity in humans: a pilot study. J Altern Complement Med. 2005 Feb;11(1):103-8. doi: 10.1089/acm.2005.11.103. PMID 15750368
- [Background] Miana L, Bastos VH, Machado S, Arias-Carrion O, Nardi AE, Almeida L, Ribeiro P, Machado D, King H, Silva JG. Changes in alpha band activity associated with application of the compression of fourth ventricular (CV-4) osteopathic procedure: a qEEG pilot study. J Bodyw Mov Ther. 2013 Jul;17(3):291-6. doi: 10.1016/j.jbmt.2012.10.002. Epub 2012 Nov 16. PMID 23768271
- [Background] Li QQ, Shi GX, Xu Q, Wang J, Liu CZ, Wang LP. Acupuncture effect and central autonomic regulation. Evid Based Complement Alternat Med. 2013;2013:267959. doi: 10.1155/2013/267959. Epub 2013 May 26. PMID 23762116
- [Background] Ahn AC, Colbert AP, Anderson BJ, Martinsen OG, Hammerschlag R, Cina S, Wayne PM, Langevin HM. Electrical properties of acupuncture points and meridians: a systematic review. Bioelectromagnetics. 2008 May;29(4):245-56. doi: 10.1002/bem.20403. PMID 18240287
- [Background] Muehsam D, Chevalier G, Barsotti T, Gurfein BT. An Overview of Biofield Devices. Glob Adv Health Med. 2015 Nov;4(Suppl):42-51. doi: 10.7453/gahmj.2015.022.suppl. Epub 2015 Nov 1. PMID 26665041
- [Background] Comunetti A, Laage S, Schiessl N, Kistler A. Characterisation of human skin conductance at acupuncture points. Experientia. 1995 Apr 15;51(4):328-31. doi: 10.1007/BF01928888. PMID 7729497
- [Background] Ahn AC, Wu J, Badger GJ, Hammerschlag R, Langevin HM. Electrical impedance along connective tissue planes associated with acupuncture meridians. BMC Complement Altern Med. 2005 May 9;5:10. doi: 10.1186/1472-6882-5-10. PMID 15882468
- [Background] Kramer S, Winterhalter K, Schober G, Becker U, Wiegele B, Kutz DF, Kolb FP, Zaps D, Lang PM, Irnich D. Characteristics of electrical skin resistance at acupuncture points in healthy humans. J Altern Complement Med. 2009 May;15(5):495-500. doi: 10.1089/acm.2008.0331. PMID 19422323
- [Background] Colbert AP, Hammerschlag R, Aickin M, McNames J. Reliability of the Prognos electrodermal device for measurements of electrical skin resistance at acupuncture points. J Altern Complement Med. 2004 Aug;10(4):610-6. doi: 10.1089/acm.2004.10.610. PMID 15353016